CLINICAL TRIAL: NCT06565871
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Phase II Study to Evaluate the Efficacy and Safety of HRS9531 Injection in Obese Subjects With Obstructive Sleep Apnea (OSA)
Brief Title: A Study of HRS9531 Injection in Obese Subjects With Obstructive Sleep Apnea
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS9531-206
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Weight Management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HRS9531 Injection low dose (Experimental)
  Interventions: Drug: HRS9531 Injection
- HRS9531 Injection high dose (Experimental)
  Interventions: Drug: HRS9531 Injection
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Injection

INTERVENTIONS:
Drug: HRS9531 Injection — Titration administration, SC
  Arms: HRS9531 Injection low dose
Drug: HRS9531 Injection — Titration administration, SC
  Arms: HRS9531 Injection high dose
Drug: Placebo Injection — SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect and safety of HRS9531 Injection in Obese Subjects with Obstructive Sleep Apnea

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age 18-65(both inclusive) at the time of signing informed consent.
2. At screening visit, BMI 24-42kg/m2(both inclusive)
3. Self-reported Diet and exercise control for at least 3 months before screening visit, and less than 5 kg self-reported change within the last 3 months.
4. At screening visit, AHI ≥15 and Obstructive Sleep Apnea on PSG

Exclusion Criteria:

1. Endocrine disorders that may significantly affect body weight, or obesity or hereditary obesity syndrome due to a single gene mutation;
2. Diabetes (except gestational diabetes)
3. There are diseases that may require systemic glucocorticoid therapy during the study period
4. Any previous or planned surgery for sleep apnea or major ear, nose or throat surgery, including tonsillectomy and adenoidectomy that still may affect breathing at time of screening Visit .Inclusion of a participant with more minor ear, nose or throat surgery (for example, deviated septum) will be at the investigator's discretion.
5. Previous or known history or family history of medullary thyroid carcinoma (MTC) or multiple endocrine adenomatosis type 2 (MEN2)
6. In or suspected of depression, bipolar disorder, suicidal tendencies, schizophrenia or other more serious mental illness;
7. Use of drugs or treatments that may lead to significant weight gain or loss within 3 months, use of stimulants and hypnotics, mirtazapine, opioids, trazodone within 3 months;
8. Patients with a history of blood donation or blood loss ≥400 ml within 3 months prior to screening, or receiving blood transfusions within 3 months
9. During the screening or before randomization ,laboratory examination meets the following conditions:

Fasting blood glucose ≥7.0 mmol/L, or HbA1c ≥6.5%; Hemoglobin <100 g/L; Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3× upper limit of normal range (ULN), total bilirubin (TBIL) ≥2.0×ULN; Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 (calculated based on serum creatinine using CKD-EPI formula); Fasting triglyceride (TG) >5.64 mmol/L (500 mg/dl); calcitonin ≥50 ng/L; Blood amylase or lipase ≥3×ULN; Thyroid stimulating hormone (TSH) <0.4 or >6.0 mIU/L; Abnormalities in other laboratory tests that the investigator determines may affect the assessment of efficacy or safety;

10、The 12-lead electrocardiogram (ECG) examination revealed clinically significant abnormalities that the investigators determined may affect the safety of the subject and QTcF>450 ms; 11、Poor blood pressure control: systolic blood pressure ≥160 mmHg, or diastolic blood pressure ≥110 mmHg, or diastolic blood pressure ≥100mmHg and deemed unsuitable for study by investigator; 12、Clinically relevant medical behavior or psychiatric disorder (other than OSA), that is associated with insomnia or excessive sleepiness in the past and at the time of screening; 13、Severe infection, severe trauma, or major or large surgery within 1 month prior to screening 14、Malignancy of any organ system within 5 years, regardless of evidence of local recurrence or metastasis; 15、A known or suspected history of alcohol and/or drug abuse; 16、The presence of a serious hematological disorder; 17、Surgery is planned during the trial (except for minor surgery that the investigators believe will not affect the trial) 18、Mentally incapacitated or speech-impaired subjects are unable to fully understand or participate in the test process; 19、In the investigator's judgment, there are circumstances (medical, psychological, social, or geographical factors, etc.) that affect subject safety or any other conditions that interfere with the evaluation of test results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in body weight | Baseline,32week

SECONDARY OUTCOMES:
Change from Baseline in Apnea-Hypopnea Index (AHI) | Baseline,32week
Proportion of subjects with weight loss of ≥5% from baseline after 32 weeks of treatment | Week 32
Proportion of subjects with weight loss of ≥10% from baseline after 32 weeks of treatment | Week 32
Proportion of subjects with weight loss of ≥15%from baseline after 32 weeks of treatment | Week 32
Change from Baseline in Body weight | Baseline,32week
Change from Baseline in BMI | Baseline,32week
Percentage change from baseline in AHI | Baseline,32week

IPD SHARING:
Plan to Share IPD: Undecided